CLINICAL TRIAL: NCT02502838
Title: The Effect of an Additional TVT on OAB Symptoms in Surgical Repair of Pelvic Organ Prolapse
Brief Title: The Effect of an Additional Stress Incontinence Procedure on Overactive Bladder During Pelvic Organ Prolapse Repair
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 15-0394
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Overactive Bladder; Pelvic Organ Prolapse
Keywords: overactive bladder; pelvic organ prolapse; TVT
MeSH Terms: conditions — Urinary Bladder, Overactive; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prolapse surgery without TVT: Patients who plan to undergo prolapse repair alone
- Prolapse surgery with TVT: Patients who plan to undergo prolapse repair with an additional TVT procedure

SUMMARY:
Pelvic organ prolapse (POP) is a common condition in women. Approximately 20% of women undergo surgical correction for POP in their lifetime. Overactive bladder symptoms (OAB) are often associated with POP in 25-69% of patients and POP has been shown to be an independent risk factor for OAB. There is scientific evidence that surgical repair of POP reduces or eliminates OAB in >85%. In addition, stress urinary incontinence (SUI) is also often associated with POP, either clinically evident or as a potential post-operative complication.

The clinical decision as to include a surgical technique to treat SUI when repairing POP surgically is still a matter of controversy. Most surgeons at the institution will include an extra procedure, specifically a retropubic sling, if SUI is clinically evident. Some will not include it unless there is urodynamic or clinical evidence of potential SUI post-operatively. Finally, some will include it regardless of clinical or urodynamic findings based on the apparent high incidence of such SUI after prolapse repair. The Tension-Free-Vaginal Tape (TVT) has been observed to reduce OAB as well as produce de-novo OAB symptoms, so the effect of TVT on OAB is still unclear.

The purpose of this study is to determine the effect of additional TVT surgery on OAB symptoms in patients undergoing POP repair. It is hoped that such data will better determine the effect of either surgical intervention strategy on OAB symptoms. This is a prospective cohort study comparing patients with OAB that undergo surgical repair of their prolapse with or without additional TVT surgery. The outcomes will be measured using pre- and post-operative validated questionnaires (PFDI-20, OAB-q short form).

DETAILED DESCRIPTION:
Hypothesis: Based on the limited data available, the investigators expect to find that there will be less improvement in OAB symptoms in women undergoing POP surgery with TVT than those undergoing POP surgery alone.

Primary Aim: To determine what effect the addition of a TVT will have on OAB symptoms in women undergoing surgical repair of pelvic organ prolapse using validated questionnaires.

Secondary Aims: To compare postoperative complications between those undergoing prolapse surgery alone and those undergoing prolapse surgery and TVT. Lastly the investigators would like to evaluate comorbidities and potential association to the degree of OAB symptoms

Methods:

Potential eligible subjects will be recruited using information provided by urogynecology staff and by reviewing the upcoming OR schedule. After subjects have been identified, the surgeon will be contacted to confirm whether or not their patient can be contacted by the research team. Only after permission has been communicated from the surgeon to the research team will the team approach the patient about potential participation.

After the patient is consented to participate she will be asked to fill out a PFDI-20 questionnaire. This is a validated questionnaire divided into 3 sections relating to prolapse symptoms, bowel symptoms and urinary symptoms, respectively. It is based on a 5 point scale- 0 for no, and then in terms of how bothersome symptoms are 2- not at all, 3- somewhat, 4- moderately, 5- quite a bit. A higher score indicates greater degree of bother. Focus will be on the UDI-6 section, pertaining to urinary symptoms.

The questions that will determine inclusion or exclusion of the patients are questions 15 and 16: "Do you usually experience frequent urination" and "Do you usually experience urine leakage associated with a feeling of urgency; that is, a strong sensation of needing to go to the bathroom?" Those who respond negatively to these questions will be excluded and those who respond affirmatively to both questions will be included.

The patients with OAB symptoms will be asked to fill out the OAB-q short form validated questionnaire which includes a 6-item symptoms bother scale (OAB-q ss) and a 13-item HRQL scale (OAB-q HRQL). This should be completed pre-operatively and then again 6 weeks, 6 months and 12 months post-operatively.

Interventions: No interventions will be made. This is an observational study.

Outcomes Primary: The primary outcome will be measured using pre- and post-operative validated questionnaires (PFDI-20, OAB-q short form). The primary study endpoint will be the Overactive Bladder Questionnaire Symptom Severity (OAB-q ss) change score 6 weeks after surgery. The change score is the score pre-operatively minus the score post-operatively. A positive score indicates lesser symptoms severity after surgery. The investigators will define a significant improvement to be a change score on the OAB-q ss≥10 based on previous work that determined that the minimally important difference in the OAB-q ss is 10 or higher.

Secondary: The secondary study endpoints will be the OAB-q HRQL change score and the UDI-6 change score calculated using the same method above.

ELIGIBILITY:
Inclusion Criteria:

* Women >21 years old with stage 2 or greater pelvic organ prolapse who plan to undergo anterior and/or apical prolapse repair
* Women who respond affirmatively to questions 15 and 16 on the PFDI-20 questionnaire
* Women with negative urine culture pre-operatively
* Women able to provide informed consent

Exclusion Criteria:

* Women with pelvic organ prolapse that respond negatively to questions 15 and 16 on the PFDI-20 questionnaire
* Women with previous urogynecologic surgery including prior hysterectomy with any type of apical support known to the patient (history of hysterectomy alone may be included)
* Women who report UTI within 1 month of recruitment (with confirmation of positive culture)
* Women with history of diagnosis of interstitial cystitis or any treatment for interstitial cystitis
* Women who undergo TVT-O (transobturator) and not retropubic TVT
* Women who undergo posterior compartment repair only
* Women who are pregnant and up to 6 weeks postpartum
* Women who undergo prolapse repair with transvaginal mesh

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present to urogynecologist for surgical management
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder Questionnaire (OAB-q short form) | baseline and 6 weeks
  Change in the OAB-q score at 6 weeks as compared to baseline. The OAB-q short form is a validated questionnaire which includes a 6-item symptoms bother scale (OAB-q ss) and a 13-item HRQL scale (OAB-q HRQL)
Overactive Bladder Questionnaire (OAB-q short form) | baseline and 6 months
  Change in the OAB-q score at 6 months as compared to baseline.
Overactive Bladder Questionnaire (OAB-q short form) | baseline and 12 months
  Change in the OAB-q score at 12 months as compared to baseline.

SECONDARY OUTCOMES:
UDI-6 change score | baseline and 6 weeks
  Change in the UDI-6 score at 6 weeks as compared to baseline. UDI-6 is a validated questionnaire pertaining to urinary symptoms. It is based on a 5 point scale- 0 for no, and then in terms of how bothersome symptoms are 2- not at all, 3- somewhat, 4- moderately, 5- quite a bit.
UDI-6 change score | baseline and 6 months
  Change in the UDI-6 score at 6 months as compared to baseline.
UDI-6 change score | baseline and 12 months
  Change in the UDI-6 score at 12 months as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States